CLINICAL TRIAL: NCT01240603
Title: Plasmodium Falciparum Clearance Rates in Response to Artesunate in Eastern Cambodia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911017; 11-I-N017
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-09-11

CONDITIONS: Malaria
Keywords: Artemisinin; Malaria; Drug Resistance; Hemoglobin E
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Plasmodium falciparum parasite clearance rates (PCRs) after oral artesunate treatment of patients with uncomplicated malaria were recently found to be significantly slower in Pailin (Western Cambodia) compared to Wang Pha (Eastern Thailand). This difference in PCRs has been attributed to different histories of artesunate drug pressure in the two areas. In Pailin, artesunate monotherapy has been used inappropriately for 30 years and is hypothesized to have selected for artemisinin-resistant parasites (slow PCRs). To investigate the potential contribution of human factors to the artemisinin resistance phenotype, we have identified a study site in Eastern Cambodia where artemisinin-resistant parasites are not believed to be present. The main aims of this study are to 1) determine whether the artemisinin resistance phenotype (i.e., a half-life longer than the 2-hour half-life observed in Wang Pha) is present in Eastern Cambodia, 2) determine whether hemoglobin E affects parasite clearance rates in vivo, 3) determine whether age-associated acquired immunity affects parasite clearance rates in vivo, and 4) identify parasite-heritable traits that are associated with slow parasite clearance rates in vivo. To meet these aims, we are conducting a prospective, longitudinal study to recruit Cambodian residents of Lumphat District in Ratanakiri Province who complain of fever and/or symptoms of malaria. Patients diagnosed with uncomplicated malaria will be treated with weight-based doses of artesunate given orally each day for 3 days followed by mefloquine given orally for 2 days. During this time, finger prick blood smears will be obtained every 6 hours until parasite density is zero. From these data, we will estimate parasite clearance rates using a half-life parameter. We will also collect parasitized red blood cell samples from malaria patients prior to antimalarial drug administration. These parasites will be tested in short-term in vitro culture experiments to determine their susceptibility to artemisinins and other antimalarial drugs.

DETAILED DESCRIPTION:
Plasmodium falciparum parasite clearance rates (PCRs) after oral artesunate treatment of patients with uncomplicated malaria were recently found to be significantly slower in Pailin (Western Cambodia) compared to Wang Pha (Eastern Thailand). This difference in PCRs has been attributed to different histories of artesunate drug pressure in the two areas. In Pailin, artesunate monotherapy has been used inappropriately for 30 years and is hypothesized to have selected for artemisinin-resistant parasites (slow PCRs). To investigate the potential contribution of human factors to the artemisinin resistance phenotype, we have identified a study site in Eastern Cambodia where artemisinin-resistant parasites are not believed to be present. The main aims of this study are to 1) determine whether the artemisinin resistance phenotype (i.e., a half-life longer than the 2-hour half-life observed in Wang Pha) is present in Eastern Cambodia, 2) determine whether hemoglobin E affects parasite clearance rates in vivo, 3) determine whether age-associated acquired immunity affects parasite clearance rates in vivo, and 4) identify parasite-heritable traits that are associated with slow parasite clearance rates in vivo. To meet these aims, we are conducting a prospective, longitudinal study to recruit Cambodian residents of Lumphat District in Ratanakiri Province who complain of fever and/or symptoms of malaria. Patients diagnosed with uncomplicated malaria will be treated with weight-based doses of artesunate given orally each day for 3 days followed by mefloquine given orally for 2 days. During this time, finger prick blood smears will be obtained every 6 hours until parasite density is zero. From these data, we will estimate parasite clearance rates using a half-life parameter. We will also collect parasitized red blood cell samples from malaria patients prior to antimalarial drug administration. These parasites will be tested in short-term in vitro culture experiments to determine their susceptibility to artemisinins and other antimalarial drugs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 2 to 65 years, inclusive

Uncomplicated P. falciparum malaria.

Tympanic temperature greater than or equal to 37.5 degree C or history of fever within the last 24 h.

P. calciparum asexual parasite density 10,000 200,000/microL, Inclusive.

Willingness to allow the storage of blood samples collected as part of the study.

Willingness and ability of the patient/guardians to comply with the protocol for the duration of the study.

EXCLUSION CRITERIA:

Severe malaria: diminished consciousness, respiratory distress, severe prostration, anuria, jaundice, hemoglobinuria, repetitive vomiting, or cessation of eating and drinking.

Non-malaria etiology of febrile illness (e.g., respiratory tract infection) evident on clinical examination.

Hematocrit < 25 percent

Treatment of present symptoms with an artemisinin compound or artemisinin-based combination therapy within the previous 7 days.

Pregnancy or breastfeeding

History or allergy or known contraindication to artemisinins or piperaquine

Splenectomy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2010-10-24; Study Completion 2013-09-11

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Center for Parasitology, Entomology, and Malaria Controk, Ministry of H, Phnom Penh, Cambodia